CLINICAL TRIAL: NCT01861535
Title: Primary Imiquimod Treatment Versus Surgery for Vulvar Intraepithelial Neoplasia
Acronym: PITVIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Austrian Science Fund (FWF) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KLI293
Record Dates: First submitted 2013-05-06; First posted 2013-05-23 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Vulvar Intraepithelial Neoplasia
Keywords: VIN; Imiquimod; Surgery; HPV; Patient satisfaction
MeSH Terms: conditions — Patient Satisfaction | interventions — Imiquimod; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Primary Imiquimod (Experimental): Treatment with imiquimod will be patient self-administered for a period of 4 months with possible extension to 6 months. A thin layer of imiquimod cream should be applied to the lesion and remain overnight without a cover. Application will be once a week for 2 weeks, then twice a week the following 2 weeks and, if tolerated, 3 times a week for the last weeks. In case of severe side-effects the number of applications can be reduced; a treatment-free period of no more than 1 week is permitted
  Interventions: Drug: Imiquimod
- Primary surgery (Active Comparator): The type of surgery (excision or ablation) will be based on clinical findings and surgeon's judgement. After excision the specimen will be histologically analyzed to assess resection margins and rule out invasion.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Drug: Imiquimod
  Other Names: Aldara
  Arms: Primary Imiquimod
Procedure: Surgery
  Other Names: Excision; Ablation
  Arms: Primary surgery

SUMMARY:
To evaluate the efficacy (defined as complete clinical response at 6 months) of imiquimod vs. standard treatment (surgery) for vulvar intraepithelial neoplasia (VIN).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed VIN (only usual type, formerly VIN 2-3)
* Visible, measurable lesion(s)
* Contraception (for premenopausal women)

Exclusion Criteria:

* Evidence of invasion
* History of cancer or severe inflammatory dermatosis of the vulva
* Pregnancy, lactation
* Immunodeficiency
* Any treatment for VIN within the previous three months
* Known hypersensitivity to imiquimod

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-06; Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Complete clinical response | 6 months
  No clinical evidence of vulvar lesion, i.e. 100% reduction of primary lesion size

SECONDARY OUTCOMES:
Clinical response/ lesion size | 6 months
  Vulvar lesions will be described, measured with calipers, mapped and photographed. The digital photos will be analyzed with a computer program (ImageJ) to calculate the total lesion size in cm². Results will be classified as: no response (NR, reduction in lesion size of 25% or less), weak partial response (wPR, 26-75% reduction), strong partial response (stPR, 76%-99% reduction) and Complete response (CR, 100% reduction).
Histologic response | 6 months
  At baseline punch biopsies will be taken from the affected areas. The site of the initial biopsy will be photodocumented to ensure that the follow-up biopsy at 6 months is taken from the same site. Histologic results will be classified as response (R): complete disappearance of usual type VIN or reduction to VIN1,or no response (NR). All biopsy samples will be analysed independently by two experienced gynecologic pathologists unaware of the treatment allocation
Extent of surgery | 6 months
  The number, types and extent of surgical procedures will be recorded. The extent of surgery will be recorded as total operated lesion size (in cm², as measured on pre-operative photograph) and relative operated lesion size (percentage of operated lesion size compared with the original pretreatment lesion size)
HPV status | 6 months
  HPV status will be measured with the qualitative cobas® HPV Test, Roche, and the the APTIMA ® HPV assay, Gen-Probe.
Clinical response/lesion size | 12 months
  Vulvar lesions will be described, measured with calipers, mapped and photographed. The digital photos will be analyzed with a computer program (ImageJ) to calculate the total lesion size in cm². Results will be classified as: no response (NR, reduction in lesion size of 25% or less), weak partial response (wPR, 26-75% reduction), strong partial response (stPR, 76%-99% reduction) and Complete response (CR, 100% reduction).
Extent of surgery | 12 months
  The number, types and extent of surgical procedures will be recorded. The extent of surgery will be recorded as total operated lesion size (in cm², as measured on pre-operative photograph) and relative operated lesion size (percentage of operated lesion size compared with the original pretreatment lesion size)
HPV status | 12 months
  HPV status will be measured with the qualitative cobas® HPV Test, Roche, and the the APTIMA ® HPV assay, Gen-Probe.

OTHER OUTCOMES:
"Cervical Dysplasia Distress" Questionnaire | 6 months
  Change from baseline in "Cervical Dysplasia Distress" score at 6 months
"Cervical Dysplasia Distress" questionnaire | 12 months
  Change from Baseline in "Cervical Dysplasia Distress" score at 12 months
"Fear of Progression" Questionnaire | 6 months
  Change from Baseline "Fear of Progression" score at 6 months.
"Fear of Progression" questionnaire | 12 months
  Change from Baseline "Fear of Progression" score at 12 months.
"Sexual activity" Questionnaire | 6 months
  Change from baseline "Sexual activity" score at 6 months
"Sexual activity" questionnaire | 12 months
  Change from baseline "Sexual activity" score at 12 months
Immune cells in the epidermis | 6 months
  Histochemical analysis of immune cells from vulvar biopsy samples will be performed at baseline and at 6 months. Frozen sections will be prepared and stained with corresponding cell markers. Immune cell populations will be quantified as number of cells per square millimetre and will be compared between the two treatment groups. The following markers and their primary antibodies will be analysed: CD1a, marker for Langerhans cells, CD94, marker for natural killer cells, CD4, marker for T-helper cells, CD8, marker for cytotoxic T-cells and CD207, marker for immature dendritic cells expressing Langerin.
Aesthetic results | 6 months
  Detailed photos of the overall vulva will be taken. Photos will be compared to photos taken at baseline and judged by 4 independent, blinded observers for aesthetic results.
Aesthetic results | 12 months
  Detailed photos of the overall vulva will be taken. Photos will be compared to photos at baseline and judged by 4 independent, blinded observers for aesthetic results.
Visual analogue scale (VAS) for assessment of pain and pruritus | 6 months
  Change of VAS score for pain and pruritus from baseline to 6 months. VAS will be assessed at baseline, 1,2 ,3,4,5 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Gerda Trutnovsky, MD, Principal Investigator — Medical University of Graz; Karl Tamussino, MD, Study Director — Medical University of Graz
Locations (9):
- Austria (9):
  - Dep. of Gynecology, Krankenhaus Barmherzige Brüder Graz, Graz, Styria
  - Dep. of Gynecology and Obstetrics, Landes Frauen- und Kinderklinik Linz, Linz, Upper Austria
  - Department of Obstetrics and Gynecology/ Medical University of Graz, Graz
  - Department of Gynecology and Obstetrics, Medical University of Innsbruck, Innsbruck
  - Dep. of Gynecology and Obstetrics, Klinikum Klagenfurt, Klagenfurt
  - Dep. of Gynecology and Obstetrics, Leoben
  - Dep. of Gynecology, Krankenhaus Barmherzige Schwestern Linz, Linz
  - Dep. of Gynecology and Obstetrics, Landeskrankenhaus Salzburg, Salzburg
  - Department of General Gynecology and Gynecology Oncology, Medical University of Vienna, Vienna

REFERENCES:
- [Derived] Muntinga CLP, de Vos van Steenwijk PJ, Kooreman LFS, Regauer S, Abdulrahman Z, Bekkers RLM, van der Burg SH, Trutnovsky G, van Esch EMG. Pre-existing infiltration with T cells and CD14+ myeloid cells is associated with treatment response to imiquimod in primary and recurrent vulvar high-grade squamous intraepithelial lesions. J Immunother Cancer. 2025 Oct 20;13(10):e012666. doi: 10.1136/jitc-2025-012666. PMID 41120128
- [Derived] Trutnovsky G, Reich O, Joura EA, Holter M, Ciresa-Konig A, Widschwendter A, Schauer C, Bogner G, Jan Z, Boandl A, Kalteis MS, Regauer S, Tamussino K. Topical imiquimod versus surgery for vulvar intraepithelial neoplasia: a multicentre, randomised, phase 3, non-inferiority trial. Lancet. 2022 May 7;399(10337):1790-1798. doi: 10.1016/S0140-6736(22)00469-X. Epub 2022 Apr 25. PMID 35483400